CLINICAL TRIAL: NCT05652660
Title: AN INTERVENTIONAL, PHASE 1, OPEN-LABEL, FIXED-SEQUENCE, 2-PERIOD STUDY TO EVALUATE THE EFFECT OF A SINGLE ORAL DOSE OF ARV-471 (PF-07850327) ON THE PHARMACOKINETICS OF ROSUVASTATIN IN HEALTHY PARTICIPANTS
Brief Title: A Study to Understand the Effect of a Study Medicine Called ARV-471 on Rosuvastatin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4891029
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin with/without ARV-471 (Experimental): Rosuvastatin administered as a single dose in Period 1 and Period 2. ARV-471 administered as a single dose in Period 2.
  Interventions: Drug: ARV-471; Drug: Rosuvastatin

INTERVENTIONS:
Drug: ARV-471 — Experimental
  Other Names: PF-07850327
Drug: Rosuvastatin — Probe substrate
  Other Names: CRESTOR®

SUMMARY:
The purpose of this study is to understand if ARV-471 affects how a BCRP substrate (rosuvastatin) gets into the body in healthy adults.

All participants in this study will receive one dose of rosuvastatin alone by mouth in Period 1. In Period 2, everyone will receive one dose of ARV-471 by mouth 90 min before one dose of rosuvastatin by mouth. The levels of rosuvastatin in Period 1 will be compared to the levels of rosuvastatin in Period 2 to determine if ARV-471 affects how rosuvastatin gets into the body differently in healthy adults.

All participants will stay at the study clinic for 10 days and 9 nights.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female participants of non-childbearing potential must be 18 to 65 years of age, inclusive at the time of signing informed consent document.
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical exam, laboratory tests, vital sign and standard 12-lead ECGs.
* BMI of 17.5 to 32 kg/m2; and a total body weight ≥45 kg.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Pregnant female participants; breastfeeding female participants; Male participants with partners currently pregnant; fertile male participants who have partners of childbearing potential and are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 90 days after the last dose of investigational product.
* Participants with known history of hypersensitivity to statin medication, sensitivity to ARV-471 or rosuvastatin or any of the formulation components of ARV-471 or rosuvastatin.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test.
* History of use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891029

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 Periods in a single fixed sequence. A total of 12 participants were enrolled in the study and received study intervention.
Groups:
- All Participants: Participants received a single oral dose of rosuvastatin 10 milligram (mg) on Period 1 Day 1. A minimum washout period of 5 days was required after rosuvastatin administration in Period 1. After completion of Period 1, participants received a single oral dose of ARV-471 (PF-07850327) 200 mg followed by a single oral dose of rosuvastatin 10 mg on Period 2 Day 1.
Period: Period 1 (5 Days)
Arm/Group | All Participants
Started | 12
Treated | 12
Completed | 12
Not Completed | 0
Period: Period 2 (4 Days)
Arm/Group | All Participants
Started | 12
Treated | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population defined as all participants enrolled and who took at least 1 dose of study intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Rosuvastatin
Description: Cmax was defined as maximum plasma concentration. Cmax of rosuvastatin was observed directly from data.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours post dose on Day 1 in Periods 1 and 2
Population: All participants enrolled and who took at least 1 dose of study intervention and had at least 1 PK parameter of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Period 1: Rosuvastatin: In Period 1 Day 1, participants received a single oral dose of rosuvastatin 10 mg.
- Period 2: ARV-471 + Rosuvastatin: In Period 2, participants received a single oral dose of ARV-471 (PF-07850327) 200 mg on Day 1 followed by a single oral dose of rosuvastatin 10 mg.
Arm/Group | Period 1: Rosuvastatin | Period 2: ARV-471 + Rosuvastatin
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 2.178 (53) | 2.625 (48)
Statistical Analysis 1: Comparison: Period 1: Rosuvastatin vs Period 2: ARV-471 + Rosuvastatin; Rosuvastatin administered alone as the Reference and ARV-471 coadministered with rosuvastatin as the Test. Natural log transformed Cmax was analyzed using a mixed effect model with treatment as fixed effects and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 120.50, 90% CI 2-sided [104.77 to 138.59] — The ratios (and 90% CIs) are expressed as percentages

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Rosuvastatin
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast of rosuvastatin was determined using Linear/Log trapezoidal method.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours post dose on Day 1 in Periods 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Period 2: ARV-471 + Rosuvastatin: In Period 2, participants received a single oral dose of ARV-471 200 mg on Day 1 followed by a single oral dose of rosuvastatin 10 mg.
Arm/Group | Period 1: Rosuvastatin | Period 2: ARV-471 + Rosuvastatin
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 31.40 (40) | 34.71 (40)
Statistical Analysis 1: Comparison: Period 1: Rosuvastatin vs Period 2: ARV-471 + Rosuvastatin; Rosuvastatin administered alone as the Reference and ARV-471 coadministered with rosuvastatin as the Test. Natural log transformed AUClast was analyzed using a mixed effect model with treatment as fixed effects and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 110.56, 90% CI 2-sided [103.53 to 118.06] — The ratios (and 90% CIs) are expressed as percentages

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship with the study intervention. SAE is defined as one of the following: is fatal or life threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE is defined as an AE with onset date occurring during the on-treatment period. AEs include all SAEs and non-SAEs.
Time Frame: From the first dose (Day 1) up to 35 days after the last dose (Day 6) of study intervention (up to 41 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Rosuvastatin | Period 2: ARV-471 + Rosuvastatin
Number analyzed (Participants) | 12 | 12
Participants
  Treatment-emergent AEs | 1 | 3
  Treatment-emergent SAEs | 0 | 0

4. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid, cystatinC); electrolytes (sodium, potassium, chloride, calcium, bicarbonate); clinical chemistry (glucose); urinalysis (dipstick [decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, bilirubin], microscopy. Abnormality was determined at the investigator's discretion.
Time Frame: Baseline (Period 1 Day -1) up to Period 2 Day 4 (10 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Rosuvastatin | Period 2: ARV-471 + Rosuvastatin
Number analyzed (Participants) | 12 | 12
Participants | 2 | 4

5. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria include a) a postdose QTc corrected using Fridericia's formula (QTcF) increased by >60 millisecond (ms) from the baseline and the absolute QTcF value >450 ms; or b) an absolute QTcF value >500 ms for any scheduled ECG.
Time Frame: Baseline (Period 1 Day 1) up to Period 2 Day 4 (9 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Rosuvastatin | Period 2: ARV-471 + Rosuvastatin
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs (blood pressure and pulse rate) were obtained with participant following at least a 5-minute rest in a supine position. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline (Period 1 Day 1) up to Period 2 Day 4 (9 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Rosuvastatin | Period 2: ARV-471 + Rosuvastatin
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose (Day 1) up to 35 days after the last dose (Day 6) of study intervention (up to 41 days)
Arm/Group | Period 1: Rosuvastatin | Period 2: ARV-471 + Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Rosuvastatin (N=12) | Period 2: ARV-471 + Rosuvastatin (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT05652660/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT05652660/SAP_001.pdf